CLINICAL TRIAL: NCT03415776
Title: Twice-Against Thrice-weekly Hemodialysis: the TATH Trial
Brief Title: Twice Against Thrice-weekly Hemodialysis
Acronym: TATH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow recruitment due to many challenges: 1-COVID-19 pandemic 2-Several units did not include their patients, 3-Many nephrologists left the country, 4-Severe economic crisis
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mabel Aoun, Dr Mabel Aoun. Head of the Department of Nephrology, Saint-Georges Hospital Ajaltoun, Saint-Joseph University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TATH2018
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; Sessions frequency; Mortality; Morbidity
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice weekly (Experimental): Two sessions of hemodialysis per week
  Interventions: Procedure: Hemodialysis
- Thrice weekly (Experimental): Three sessions of hemodialysis per week
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: Hemodialysis — Renal replacement therapy

SUMMARY:
Hemodialysis is the most worldwide prescribed renal replacement therapy for patients with end-stage renal disease. The frequency of sessions per week remains a debatable issue. In the majority of developed Western and Asian countries, patients on chronic hemodialysis are undergoing three dialysis sessions weekly. In developing countries and some developed countries, a twice-weekly schedule independent of residual kidney function is still accepted, sometimes because of lack of resources and some other times because of patients' resistance to undergo three sessions per week. The primary objective of this trial is to assess the total mortality of patients on thrice against twice-weekly hemodialysis. The secondary objectives are a) to compare the rate of urgent supplementary hemodialysis sessions between the two arms, mainly those due to pulmonary edema and hyperkalemia, b) to compare the number of hospitalizations and duration of stay, c) to compare the rate of uncontrolled hypertension between the two groups, d) to analyze the quantity of erythropoiesis-stimulating agents (ESAs) in units to achieve a haemoglobin (Hb) 11 to 11.5 g/dl, e) to assess the factors associated with a higher mortality in the two groups.

DETAILED DESCRIPTION:
Hemodialysis (HD) is the most worldwide prescribed renal replacement therapy for patients with end-stage renal disease. This treatment that relies heavily on technology has undergone major modifications in the last five decades in order to improve patients' outcomes. Those changes that aimed at reducing the morbidity and mortality of patients targeted mainly the water purification system, the membrane's permeability and biocompatibility, the dialysate composition and the dose of hemodialysis. However, the frequency of sessions per week remains a debatable issue influenced by the fluctuating scientific evidence and the patient's disapproval of being increasingly dependent on a machine.

In the majority of developed Western and Asian countries, patients on chronic hemodialysis are undergoing three dialysis sessions weekly.

In 2007 the European guidelines recommended the thrice-weekly hemodialysis with a session duration 3-5 hours. This dose of treatment will ensure hemodialysis sessions adequacy defined as urea reduction ratio >65% . However thrice-weekly hemodialysis has been established worldwide without randomized clinical trials. The rationale behind the thrice-weekly dialysis seems to be the uncertainty about dialysis adequacy and the risk of malnutrition, anemia and intra-dialytic hypotension with twice-weekly sessions. Several cohorts have also shown a favorable effect on survival with thrice compared to twice-weekly hemodialysis especially when duration of treatment per week of the twice-weekly schedule was less than 8 hours.

Incremental hemodialysis is defined as starting dialysis twice weekly for those who have a substantial renal urea clearance and switching after 3 months to three times weekly. A large retrospective study from the US showed that incremental hemodialysis compared to conventional hemodialysis (three times per week) improved mortality in those with a renal urea clearance >=3 ml/min/1.73 m2 or urine volume > 600 ml/day. The rationale behind the incremental schedule is that preserving residual kidney function would lead to better outcomes. However based on this incremental method, patients should be watched closely for the residual kidney function and switched at the right moment to three sessions per week otherwise there will be an overlap between the two phases and an information bias regarding the timing of residual renal function loss.

In developing countries and some developed countries, a twice-weekly schedule independent of residual kidney function is still accepted, sometimes because of lack of resources and some other times because of patients' resistance to undergo three sessions per week. Several studies have shown that patients on twice-weekly hemodialysis without residual kidney function have a shorter survival than those on three times per week. A recent prospective study from Korea showed that residual kidney function is not the only factor that would favor thrice over twice weekly HD. Another retrospective Indian study showed similar mortality between those on twice versus thrice-weekly HD while a Chinese observational study demonstrated longer survival in anuric patients on twice- than thrice-weekly dialysis. All these controversial studies make it unclear whether patients are still allowed to undergo twice-weekly hemodialysis.

Lebanon is a developing upper middle-income country from the Eastern Mediterranean region where around 3800 patients are undergoing chronic hemodialysis three or twice weekly. Although the Lebanese Ministry of Public Health recommended in 2014 that all patients on chronic hemodialysis be dialyzed three times weekly, many nephrologists are still allowing the twice schedule if it is more convenient to the patients. With these circumstances, Lebanon appears an attractive place to study the difference in outcomes between the two hemodialysis schedules.

Trial design This is a non-randomized, multicenter, clinical trial. Randomization was considered unethical and contradictory with the current international guidelines. Therefore patient's allocation was left at the nephrologist and patient's agreement.

Crossover will be allowed during follow-up to limit attrition. This study will assess the equivalence between the two schedules.

Methods: participants, interventions and outcomes

Study setting Hemodialysis patients will be recruited from multiple Lebanese HD centers. Lebanon is divided into 9 governorates and includes 77 HD units. From each governorate 50% of the units will participate in the trial.

Interventions Patients will be assigned to one of two groups upon their agreement with the treating nephrologist: Group 1 will receive three sessions of hemodialysis weekly. Group 2 will receive two sessions weekly.

Participant timeline Recruitment of patients will be done over two years or until the pre-determined sample size is reached whichever comes earlier.

Sample size Knowing that the proportion of death varies between 10% and 40%, if we consider a two sided alpha of 5%, a power of 80% and a small effect size = 0.20 (Cohen's d), the total sample size needed would be 806 patients. Assuming an attrition rate of 10%, we would need 806/0.9 = 896 patients. The representative sample size for this study is ~900 patients. 600 patients are necessary for the three times weekly arm and 300 patients for the twice weekly arm.

Recruitment It may be difficult to reach 300 patients on twice weekly so the recruitment will go on till this number is reached.

Methods: Data collection, management, and analysis

Data collection methods eCRF (electronic case report form) will be used for data capture. Data for demographics, comorbidities, laboratory results, medications and dialysis prescription will be collected from the patients' medical records at dialysis initiation.

The following variables will be studied:

Baseline characteristics: age, gender, body mass index (BMI), diabetes, smoking, hypertension, hyperlipidemia, cause of end-stage renal disease (ESRD), previous cardiovascular disease, atrial fibrillation, dementia, Laboratory: serum creatinine (with corresponding estimated glomerular filtration rate (eGFR), phosphate, calcium, albumin, potassium, sodium, bicarbonate, hemoglobin, parathyroid hormone (PTH), alkaline phosphatase, ferritin, transferrin saturation, uric acid, hepatitis B (HBV) and hepatitis C (HCV) serologies.

Residual renal function: Urine volume and renal urea clearance will be assessed at baseline by collecting the 24 hour-urine at dialysis initiation.

Medications: statins, calcium-based and non-calcium-based phosphate binders, vitamin D, antihypertensive medications, antiplatelet agents, erythropoiesis stimulating agents (ESA) dose, renin-angiotensin system inhibitors, oral anticoagulants.

Dialysis prescription: Number of hours per week, blood flow, dialysate flow, type of vascular access (catheter, graft or arteriovenous fistula), filter membranes (surface, low-flux or high-flux), dialysate potassium and calcium content will be collected.

Definitions Chronic kidney disease stage 5 is defined as an eGFR <15 ml/min. Coronary artery disease is defined as a history of myocardial infarction or obstructive coronary artery disease, treated medically or interventionally. Diabetes and hypertension are defined as having a history for antidiabetic or antihypertensive treatment respectively.

Uncontrolled hypertension is defined as a pre-dialysis BP > 160/90 in more than 2/3 of the sessions. Residual kidney function is defined as a diuresis > 500 ml/d on a non-dialysis day.

Statistical analysis Continuous variables will be presented as mean ± standard deviation (SD). Differences between the study groups will be tested using χ2 tests (for categorical variables). Bivariate correlation analysis will be performed using the Pearson's correlation coefficient. The Kaplan-Meier method will be used to estimate the cumulative survival. Cox regression will be used to determine the effect of dialysis frequency and other covariates on mortality. Analysis will be performed on an intention-to-treat basis. Statistical analysis will be performed with SPSS. A P-value of ≤0.05 will be considered statistically significant.

Methods: Monitoring

Data monitoring Follow-up with laboratory measurements and medication dosage Every month: hemoglobin, calcium, phosphorus, urea, creatinine, potassium, sodium, bicarbonate.

Every 4 months: PTH, ferritin, transferrin saturation. Every year: lipid panel, albumin. All these biological parameters will be measured with the standard laboratory techniques and medications adjusted to maintain serum calcium, phosphate and PTH within the target range.

Total ESA quantity used for each patient, as well as doses of alfacalcidol, cinacalcet, phosphate binders and antihypertensive treatment will be collected every 3 months.

Clinical follow-up Data that will be collected monthly includes: mid-week pre-dialysis systolic and diastolic blood pressure, average interdialytic fluid gain, number, causes (myocardial infarction, angina, atrial fibrillation, pulmonary edema, hyperkalemia) and length of hospital stay (LOS), residual kidney function, number of vascular access thrombosis. Blood pressure will be recorded every week and presented as a monthly average.

ELIGIBILITY:
Inclusion Criteria:

* all incident patients 18 years and older with CKD stage 5 started on hemodialysis.

Exclusion Criteria:

* late-stage cancer patients and participants who are terminally ill defined as having an expected survival of less than 3 months.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Mortality | 0-24 months
  All cause mortality

SECONDARY OUTCOMES:
Supplementary dialysis sessions | 0-12 months
  Rate of supplementary hemodialysis sessions for pulmonary oedema or hyperkalemia
Hospitalizations | 0-12 months
  Number of hospitalisations
Uncontrolled hypertension | 0-12 months
  Rate of uncontrolled hypertension, Uncontrolled hypertension is defined as a pre-dialysis BP > 160/90 in more than 2/3 of the sessions.
ESA dose | 0-12 months
  Total ESA dose administered

CONTACTS AND LOCATIONS:
Overall Officials: Mabel Aoun, MD, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint-Georges Hospital, Ajaltoun, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aoun M, Finianos S, Beaini C, Sleilaty G, Ghaleb R, Nourie N, Kais S, Hajal JE, Alameddine R, Boueri C, Ghoul BE, Zeidan S, Azar H, Dfouni A, Hawi J, Mechref Z, Hage V, Chelala D. Twice against thrice-weekly hemodialysis (TATH): a multicenter nonrandomized trial. BMC Nephrol. 2025 Apr 5;26(1):176. doi: 10.1186/s12882-025-04105-3. PMID 40188011